CLINICAL TRIAL: NCT07152782
Title: Trastuzumab Deruxtecan With or Without Neratinib for HER2-positive Unresectable and/or Metastatic Breast Cancer With Brain Metastasis: A Multicenter, Randomized, Open Label, Phase II Trial (THUNDER Trial)
Brief Title: T-DXd With or Without Neratinib for HER2 Positive Breast Cancer With Brain Metastasis
Acronym: THUNDER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC- N0101
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer With Brain Metastasis; HER2-positive Breast Cancer
Keywords: Breast Cancer with Brain Metastasis; HER2-positive Breast Cancer; Trastuzumab Deruxtecan; Neratinib
MeSH Terms: interventions — neratinib; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-DXd (Active Comparator): T-DXd: 5.4mg/kg intravenously (IV) every 3 weeks (Q3W).
  Interventions: Drug: Trastuzumab Deruxtecan
- T-DXd+Neratinib (Experimental): T-DXd: 5.4mg/kg intravenously (IV) every 3 weeks (Q3W). Neratinib: 200mg po, D1-21, every 3 weeks (Q3W).
  Interventions: Drug: Neratinib; Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Neratinib — Neratinib, as an irreversible pan-HER tyrosine kinase inhibitor (TKI), holds a unique position in the treatment of HER2-positive breast cancer. From a molecular perspective, Neratinib irreversibly binds to the intracellular kinase domains of HER1 (EGFR), HER2, and HER4 through covalent bonds, comprehensively blocking signal transduction of the HER family. This mechanism of action is markedly different from reversible TKIs such as lapatinib. Neratinib's irreversible binding characteristic allows for a more sustained inhibition of target activity, maintaining anti-tumor effects even after drug plasma concentrations have decreased. This feature is particularly important for HER2-positive breast cancer, which requires continuous suppression of proliferative signals.
  Arms: T-DXd+Neratinib
Drug: Trastuzumab Deruxtecan — Trastuzumab deruxtecan (T-DXd) is an antibody-drug conjugate (ADC) composed of an anti-HER2 monoclonal antibody (trastuzumab), a cleavable linker, and a topoisomerase I inhibitor (an exatecan derivative). It targets and binds to HER2-positive tumor cells, internalizes, and releases cytotoxic drugs to induce DNA damage and apoptosis. It also has a "bystander effect" that can kill neighboring tumor cells with low HER2 expression, enhancing anti-tumor activity. T-DXd has shown significant efficacy in HER2-positive advanced breast cancer, with key clinical trials (such as DESTINY-Breast03) confirming that its progression-free survival (PFS) and overall survival (OS) are superior to traditional second-line treatments, with a median PFS reaching 28.8 months. Additionally, for HER2-low-expressing (IHC 1+ or 2+/ISH-) metastatic breast cancer (in the DESTINY-Breast04 study), T-DXd can extend PFS and OS, becoming the first targeted therapy to alter the survival outcomes of such patients
  Other Names: DS8201

SUMMARY:
A phase II, open-label, multicenter, randomized controlled trial exploring the efficacy and safety of Trastuzumab Deruxtecan combined with or without Neratinib in HER2-positive breast cancer with brain metastasis

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open-label, Phase II, randomized controlled clinical trial aimed at evaluating the efficacy and safety of T-DXd with or without neratinib in patients with HER2-positive breast cancer with brain metastases. All eligible subjects will be randomly assigned in a 1:1 ratio across multiple centers in China to receive either T-DXd combined with neratinib or T-DXd monotherapy until extracranial progression as defined by RECIST 1.1, unless unacceptable toxicity occurs, consent is withdrawn, or other criteria for discontinuation are met.

ELIGIBILITY:
Inclusion Criteria:

-

Participants must meet all of the following inclusion criteria in order to be enrolled in this study:

1. Female, aged 18-70 years old.
2. ECOG score ranges from 0 to 1.
3. Expected survival period is greater than 12 weeks.
4. Histologically confirmed invasive HER2 positive breast cancer (HER2 IHC+++or FISH/CISH positive, all samples need to be verified by the pathology department of the research center).
5. Tumor staging: recurrent or metastatic breast cancer; Patients with local recurrence need to be confirmed by the researcher that radical surgical resection cannot be performed.
6. The subject has at least one lesion (measurable and/or unmeasurable) that has not received radiation therapy in the past.
7. MRI or CT shows brain metastasis and meets one of the following conditions:

   i) Untreated brain parenchymal metastases detected through imaging screening;

   Ii) Stable or progressive brain parenchymal metastases that have undergone previous local treatment and meet one of the following conditions:
   1. Stable imaging for ≥ 4 weeks;
   2. New brain parenchymal metastases detected by MR or CT.
8. Transfer treatment ≤ 2 lines, and did not receive T-DXd or nalatinib.
9. The main organ functions are basically normal, meeting the following conditions:

   1. The standard for blood routine examination should meet: HB ≥ 90g/L (no blood transfusion within 14 days); ANC≥1.5×109/L；PLT≥75×109/L；
   2. Biochemical tests must meet the following standards: TBIL ≤ 1.5 × ULN (upper limit of normal value); ALT and AST ≤ 3 × ULN; If there is liver metastasis, ALT and AST should be ≤ 5 × ULN; Serum Cr ≤ 1.5 × ULN, endogenous creatinine clearance rate ≥ 30mL/min (Cockcroft Gault formula).
10. Prior to enrollment, the use of mannitol and hormone therapy is allowed, but the medication dosage should be stable for at least one week without the need for an increase.
11. Female participants with fertility agreed to take effective contraceptive measures until 3 months after the last use of medication.
12. The subjects voluntarily joined this study, signed informed consent forms, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

-

Subjects with any of the following conditions are not eligible for inclusion in this study:

1. Transfer treatment exceeding 2 lines, or previous use of T-DXd or nalatinib.
2. Meningeal metastasis.
3. Brain metastases that require emergency intervention treatment, or brain metastases that require treatment with more than 3mg/d dexamethasone or equivalent drugs.
4. A history of clinically significant or uncontrolled heart disease, including congestive heart failure, angina, myocardial infarction within the past 6 months, or ventricular arrhythmia.
5. Due to ongoing grade ≥ 2 adverse reactions caused by previous treatments (excluding hair loss).
6. Pregnancy period.
7. Other malignant tumors within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin.
8. Unable to swallow, chronic diarrhea, and intestinal obstruction, there are multiple factors that affect medication intake and absorption.
9. There is a third interstitial fluid accumulation that cannot be controlled by drainage or other methods (such as a large amount of pleural fluid and ascites).
10. Participated in clinical trials of other anti-tumor drugs within 4 weeks prior to the first use of the investigational drug.
11. Long term unhealed wounds or fractures with incomplete healing.
12. Known subjects with active HBV or HCV infection.
13. Active primary immunodeficiency, known to be HIV positive.
14. Uncontrolled infections requiring intravenous injection of antibiotics, antiviral drugs, or antifungal drugs.
15. A history of non communicable ILD/pneumonia requiring steroids, currently suffering from ILD/pneumonia, or unable to rule out suspected ILD/pneumonia through imaging during screening.
16. Lung standard:

    1. Pulmonary specific comorbidities with clinically significant diseases, including but not limited to any potential pulmonary diseases (such as pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease, restrictive pulmonary disease, pleural effusion, etc. within 3 months of recruitment).
    2. Any autoimmune disease, connective tissue disease, or inflammatory disease (such as rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc.). There are records or suspicions of lung involvement during screening. For participants participating in the study, all detailed information about the disease should be recorded in the CRF.
    3. Previous complete lung resection surgery.
17. Individuals with allergies, or those with a known history of allergies to the components of this medication regimen, or subjects who are allergic to other monoclonal antibodies.

Researchers believe that substance abuse or medical conditions may interfere with participants' participation in clinical studies or the evaluation of clinical study results.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | 24 months
  Time to progressive disease (according to RECIST1.1)

SECONDARY OUTCOMES:
CNS Progression-free survival (CNS-PFS) | 24 months
  Time from enrollment to the first radiographic documented disease progression (PD) of all CNS target lesions (RANO-BM criteria) or death from any cause without progression was recorded.
Objective response rate (ORR) | 24 months
  Partial response is defined as a decrease by 30% or more in sums of longest diameter of measurable target lesions
CNS Objective response rate (CNS-ORR) | 24 months
  The proportion of patients with complete response (CR) and partial response (PR) evaluated as the best response observed from enrollment to progression of all CNS target lesions assessed according to RANO-BM criteria among the total number of patients who could be evaluated.
Overall survival (OS) | 48 months
  Time from the enrollment to death of any cause
Safety and Tolerability | 24 months
  Safety and Tolerability Will be Assessed According to Standard (CTCAE Version 5.0) Toxicity Reporting Criteria.

IPD SHARING:
Plan to Share IPD: No